CLINICAL TRIAL: NCT00003411
Title: Phase I Dose Escalation and Pharmacokinetics Study of the Radiosensitizer, Gadolinium Texaphyrin (Gd-Tex, NSC 695238) With Concurrent Radiotherapy in Advanced Biliary Tree and Pancreatic Cancers
Brief Title: Radiation Therapy in Treating Patients With Bile Duct, Gallbladder, or Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nathan Bahary, MD, Associate Professor, University of Pittsburgh
Purpose: Treatment
Other Study IDs: PCI-97-108; CDR0000066423 (Registry Identifier: PDQ (Physician Data Query)); NCI-T97-0109
Record Dates: First submitted 1999-11-01; First posted 2004-02-20 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Pancreatic Cancer
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; unresectable gallbladder cancer; unresectable extrahepatic bile duct cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Pancreatic Neoplasms | interventions — motexafin gadolinium; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: motexafin gadolinium
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Motexafin gadolinium may increase the effectiveness of radiation therapy by making tumor cells more sensitive to treatment.

PURPOSE: Phase I trial to study the effectiveness of radiation therapy plus motexafin gadolinium in treating patients with bile duct, gallbladder, or pancreatic cancer that cannot be removed surgically.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and toxicity of motexafin gadolinium (PCI-0120) when administered concurrently with radiotherapy in patients with locally advanced unresectable pancreatic or biliary tree tumors. II. Assess the pharmacokinetics of this regimen in these patients. III. Assess tumor uptake of PCI-0120 (by MRI signal characteristics) in these patients. IV. Determine the maximum tolerated dose of PCI-0120 in these patients. V. Determine the objective response (by radiologic criteria) in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of motexafin gadolinium (PCI-0120). Patients receive PCI-0120 IV over 15 minutes 3 times weekly concurrently with external beam radiotherapy (EBRT) 5 days a week for 5.5 weeks. After completion of EBRT and PCI-0120, patients may undergo radiotherapy boost for 5 consecutive days. Cohorts of 3-6 patients receive escalating doses of PCI-0120 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A total of 6-12 patients are treated at the recommended phase II dose. The recommended phase II dose is defined as the dose immediately preceding the MTD. Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 18-21 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed locally advanced, unresectable carcinoma of the biliary tree or pancreas Metastatic disease allowed on a case by case basis provided the following criteria exists: Minimal or low volume disease Need for palliative radiotherapy to primary tumor with or without motexafin gadolinium No requirement for systemic therapy Measurable disease in at least 2 dimensions No ascites requiring therapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 No history of glucose-6-phosphate dehydrogenase deficiency Hepatic: Bilirubin no greater than 2.0 mg/dL AST and ALT less than 3 times upper limit of normal Renal: Creatinine no greater than 1.6 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No history of porphyria No active infection No physical or psychological illness that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics No prior radiotherapy to primary site of tumor Surgery: See Disease Characteristics At least 3 weeks since prior major surgery Other: At least 4 weeks since prior investigational drugs No other concurrent investigational antineoplastic drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-11; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh K. Ramanathan, MD, Study Chair — University of Pittsburgh
Locations (3):
- United States (3):
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin